CLINICAL TRIAL: NCT01950702
Title: Laryngoscope Assisted Lightwand Can Provide More Successful Intubation Than Lightwand Alone in Patients With Cervical Spine Injury : A Prospective Randomized Study
Brief Title: Laryngoscope Asssited Lightwand Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: php3
Record Dates: First submitted 2013-09-11; First posted 2013-09-25 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Cervical Spine Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lightwand intubation (Active Comparator): After standard total intravenous anesthesia using propofol and remifentanil continuous infusion, traditional lightwand intubation was done by pre-specified anesthesiologist who experienced more than 100 times of lightwand intubation.
  Patient's head were fixed at neutral position during all intubation period.
  Interventions: Procedure: Lightwand intubation
- Laryngoscope assisted lightwand intubation (Experimental): After standard total intravenous anesthesia using propofol and remifentanil continuous infusion, lightwand intubation using specific device(Macintosh laryngosope, female:3/Male:4) was done by pre-specified anesthesiologist who experienced more than 100 times of laryngoscope assisted lightwand intubation.
  Interventions: Procedure: Laryngoscope assisted lightwand intubation

INTERVENTIONS:
Procedure: Laryngoscope assisted lightwand intubation — After standard monitoring(EKG, pulse oximetry, NIBP), participants were induced with remifentanil and propofol continuous infusion, using targe-controlled infusion device with prexoygenation with 100% oxygen.
  Manual in-line stabilization was applied with velcro during intubation to maintain neutral head position.
  The Macintosh laryngoscope (female: 3rd blade, male: 4th blade) was inserted into the oral cavity to provide direct view of the epiglottis and then the tip of the lightwand was placed below the epiglottis.
  Other Names: The Macintosh laryngoscope (female: 3rd blade, male: 4th blade); lightwand (Surch-Lite, Aaron Medical Industries, St. Petersburg, FL)
  Arms: Laryngoscope assisted lightwand intubation
Procedure: Lightwand intubation — After standard monitoring(EKG, pulse oximetry, NIBP), participants were induced with remifentanil and propofol continuous infusion, using targe-controlled infusion device with prexoygenation with 100% oxygen.
  Manual in-line stabilization was applied with velcro during intubation to maintain neutral head position.
  After 2min from administration of rocuronium, the clinician holds the wand similar to a pencil, stands directly behind the patient's head, inserts the device into the side of the mouth and sweeps the tip to the midline. After confirmation of precise location via clear light source on anterior neck, endotracheal tube was inserted and withdrawn lightwand.
  Other Names: Surch-Lite, Aaron Medical Industries, St. Petersburg, FL
  Arms: Lightwand intubation

SUMMARY:
To evaluate the success rate for intubation of laryngocope assisted lightwand intubation.

DETAILED DESCRIPTION:
Light wand intubation is well known for safety intubation in cervical injury patiets. Traditional method of using light wand can damage the supraglottic cavity by scooping the apparatus. The investigators try to evaluate the efficacy of laryngoscope assisted light wand intubation compared to traditional method of using light wand alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for cervical spine surgery under general anesthesia

Exclusion Criteria:

* congenital or acquired abnormalities of the upper airway, tumours, polyps, trauma, abscesses, inflammation, or foreign bodies in the upper airway
* history of gastro-esophageal reflux disease, previous airway surgery, an increased risk of aspiration, coagulation disorders
* American Society of Anesthesiologists physical status ≥ 3

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The success rate of intubation | up to 60 seconds
  confirm the success intubation via end tidal CO2 measurement

SECONDARY OUTCOMES:
lightwand search (=intubation) time | from the insertion of the lightwand or laryngoscope into the oral cavity to the point of transillumination over the cricothyroid membrane within 60 sec.
  Check the time(sec) from insertion of the lightwand or laryngoscopy into the oral cavity to push the endotracheal tube into the trachea.
The times of scooping of lightwand | within 1min after insertion of lightwand
  Within 1min after insertion of lightwand into oral cavity, check the scooping time of lightwand during intubation.

OTHER OUTCOMES:
score of postoperative sorethroat | at postanesthetic care unit (PACU) within 1hr after end of anesthesia
  check the postoperative sorethroat at PACU in each patient. Numeric rating scale(NRS) was used to measure the severity of pain 0 to 10.
Incidence of moderate to severe postoperative sorethroat | at postanesthetic care unit (PACU) within 1hr after end of anesthesia
  check the postoperative sorethroat >3 at PACU in each patient. Numeric rating scale(NRS) was used to measure the severity of pain 0 to 10. 0-3 : mild 4-7 : moderate 8-10 : severe
other possible postoperative complications | just after extubation, an expected average of 1hr
  tinged blood to endotracheal tube or in oral cavity. hoarseness

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Pyung Park, MD PhD, Study Director — Professor; Eugene Kim, MD, Principal Investigator — fellow
Locations (1):
- Seoul National University of Hospital, Seoul, Jongno-Gu, South Korea